CLINICAL TRIAL: NCT05183113
Title: Neurovascular Mechanisms of Intermittent Hypoxia Induced Neural Plasticity
Brief Title: Measuring the Neurological Benefits of Intermittent Hypoxia Therapy With MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Molly Bright, Assistant Professor; Physical Therapy and Human Movement Sciences; Feinberg School of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SP0051925
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Acute Intermittent Hypoxia; Magnetic Resonance Imaging
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acute Intermittent Hypoxia (Experimental): Both healthy participants and those with spinal cord injury will receive the acute intermittent hypoxia (AIH) intervention. All participants are imaged pre- and post-AIH intervention, and thus serve as a self-comparison to observe the hypothesized improvement in bilateral hand strength.
  Interventions: Other: Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — Participants will wear a non-rebreathing face mask and alternate between breathing 9% O2 gas mixture for up to 1 minute, or until the target SpO2 of 85 percent is reached, and normal room air (21 percent O2) until 2 minutes are complete. This cycle will be repeated 15 times, resulting in a 30-minute protocol.

SUMMARY:
This study uses Magnetic Resonance Imaging to image the brain and spinal cord before and after an Intermittent Hypoxia intervention. Acquiring these scans in patients with chronic cervical spinal cord injury and uninjured controls will enable characterization of changes in neurovascular physiology caused by this promising new therapy.

DETAILED DESCRIPTION:
Acute intermittent hypoxia (AIH) is an emerging, safe technique for facilitating neural plasticity in individuals with chronic spinal cord injury (SCI), demonstrating significant transient improvements in respiratory function, plantar flexion, locomotor function, and hand dexterity and strength. Although these studies observe some degree of success eliciting plasticity, we lack a framework for systematic optimization of the AIH protocol for individual patients.

Better understanding of what physiological mechanisms drive AIH-induced neural plasticity in humans will directly inform the development of AIH as an effective treatment option in chronic SCI. This study applies magnetic resonance imaging (MRI) to test how AIH influences vascular and neural properties of the brain and spinal cord.

Individuals with SCI and uninjured participants will be recruited to undergo two MRI scan sessions on one day. In between these scan sessions, participants will undergo a single 30-minute session of AIH. In each scan session, functional MRI will assess AIH-induced changes in neural activation patterns during motor tasks (unilateral isometric hand grasping tasks) and vascular reactivity to breath hold tasks (transient hypocapnia to induce vasodilation). Additional structural scans will be acquired to aid in image analysis.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the following inclusion criteria:

* Between the ages of 18-60 years
* Safe to be scanned using MRI
* Able to communicate in English
* Ability to sign informed consent

In addition, the participants recruited with SCI must meet the following criteria:

* History of a traumatic spinal cord injury, inclusive of levels C2-T1
* At least 6 months since onset of spinal cord injury
* Cause of the spinal cord injury was non-progressive
* Ability to complete and comply with information within the informed consent
* Ability to close and open at least one hand without assistance

Exclusion Criteria:

* MRI contraindications as indicated on MRI safety screening form
* Subjects with pacemakers, cochlear (in the ear) implants, or aneurysm clips or subjects who have worked with metal
* Women who are currently pregnant, nursing, or planning on becoming pregnant
* Individuals with severe claustrophobia
* Subjects unwilling or unable to give written informed consent in English
* Prisoners
* Frequent smokers (greater than 5 cigarettes per day)
* Blood pressure greater than 160/110 or less than 85/55.
* Individuals who report headaches, feeling dizzy or light-headed, or have heart palpitations on the day of the study.
* Diagnosis of any of the following comorbid conditions: congestive heart failure, cardiac arrhythmias, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, emphysema, severe asthma, previous myocardial infraction or known carotid/intracerebral artery stenosis, presence of active deep venous thrombosis, or cancer.
* Individuals who utilize mechanical ventilation or have a tracheostomy
* Individuals who utilize an intrathecal baclofen pump
* Orthopedic injury affecting upper extremities
* Currently participating in any other hypoxia related study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI activation in motor cortex during isometric hand grip tasks | Immediately before and ~ 1-hour after AIH on the same day
  Assess AIH-induced changes in %BOLD activation within the left and right motor cortices during unilateral isometric hand grasping tasks targeting submaximal force levels with real-time feedback.
BOLD fMRI vascular reactivity to a breath-hold task | Immediately before and ~ 1-hour after AIH on the same day
  Measurements of breath-hold induced vasodilation (vascular reactivity, in units of %BOLD/mmHg end-tidal CO2) acquired via functional MRI in the brain and spinal cord.

CONTACTS AND LOCATIONS:
Overall Officials: Molly G Bright, DPhil, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
MR imaging data and the associated physiologic data collected during MRI scanning will be shared in an anonymized format. These data will be made available to public through the Open Science Framework (osf.io) or similar public repository.
Time Frame: At time of publication (or within one year of project completion, whichever occurs first).
Access Criteria: Data will be anonymized and made publicly available, and at that time no approval is needed and therefore there are no access criteria.

REFERENCES:
- [Background] Golder FJ, Mitchell GS. Spinal synaptic enhancement with acute intermittent hypoxia improves respiratory function after chronic cervical spinal cord injury. J Neurosci. 2005 Mar 16;25(11):2925-32. doi: 10.1523/JNEUROSCI.0148-05.2005. PMID 15772352
- [Background] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Li Y, Lucas-Osma AM, Black S, Bandet MV, Stephens MJ, Vavrek R, Sanelli L, Fenrich KK, Di Narzo AF, Dracheva S, Winship IR, Fouad K, Bennett DJ. Pericytes impair capillary blood flow and motor function after chronic spinal cord injury. Nat Med. 2017 Jun;23(6):733-741. doi: 10.1038/nm.4331. Epub 2017 May 1. PMID 28459438